CLINICAL TRIAL: NCT00092859
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety, Tolerability, and Efficacy of MK0557 in Obese Patients
Brief Title: A 2-Year Study of an Investigational Drug in Obese Patients (0557-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0557-011; MK0557-011; 2004_030
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — spiro(cyclohexane-1,3'(1'H)-furo(3,4-C)pyridine)-4-carboxamide, N-(1-(2-fluorophenyl)-1h-pyrazol-3-yl)-1'-oxo-, trans-

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0557

SUMMARY:
This is a 2-year study to assess the safety, tolerability, and efficacy of an investigational drug in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Obese men and nonpregnant women at least 18 years of age with a specific body mass index (height and weight ratio) required by the study

Exclusion Criteria:

* Patients with uncontrolled high blood pressure and/or diabetes mellitus (high blood sugar)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2003-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Body weight after 1 year of treatment. Safety and tolerability for 2 years. | After 1 & 2 years of treatment

SECONDARY OUTCOMES:
Durability of weight loss over two years. | Over two years.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC